CLINICAL TRIAL: NCT00771797
Title: Clinical Study to Assess the Clinical Efficacy of Flavanol-rich Cocoa on Vascular Function in Diabetic Patients With PAOD
Brief Title: Peripheral Artery Occlusive Diseases (PAOD) Study - Clinical Assessment
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: investigator took study to university hospital duesseldorf
Sponsor: RWTH Aachen University (Other)
Collaborators: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Heinrich-Heine-University Düsseldorf, Clinic for Cardiology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PAOD Study
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Peripheral Artery Disease
Keywords: PAOD; diabetis; vascular function; in diabetics with PAOD
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Treatement with low dose flavanoids over 60 days
  Interventions: Dietary Supplement: low dose flavanoids
- 2 (Experimental): Treatment with high dose flavanoids over 60 days
  Interventions: Dietary Supplement: high dose flavanoids

INTERVENTIONS:
Dietary Supplement: high dose flavanoids — flavanoid rich cocoa 2 times daily over 60 days
  Arms: 2
Dietary Supplement: low dose flavanoids — treatment with flavanoid-low cocoa two times daily over 60 days
  Arms: 1

SUMMARY:
To assess the clinical efficacy and to simultaneously explore the underlying molecular mechanisms of the beneficial effects of flavanol-rich cocoa on vascular function diabetic patients with peripheral artery occlusive diseases (PAOD) of the lower extremities will be investigated.

DETAILED DESCRIPTION:
50 Type 2 diabetics according to the criteria of the American Diabetes Association suffering from PAOD with a pain free walking distance less than 200 m will be enrolled. In a randomized controlled parallel group study the before established novel 5-level approach of vascular diagnostics will be realised. In order to test the hypothesis, whether cocoa rich in flavanols improves vascular function of diabetic PAOD subjects will regularly intake flavanol rich cocoa (group 1: 975 mg/d, n=50 versus group 2: 90 mg/d, n=50) over a period of two months. Clinical endpoints are the Ankle-Brachial-Index, measured by Doppler ultrasound and the pain-free walking distance determined by a treadmill ergometer. All parameters of vascular diagnostic (see 5-level approach above) will be determined before and two month after cocoa ingestion.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetes mellitus type 2 defined by the criteria of the American Diabetes Association

   * Fasted plasma glucose greater than 126 mg/dL
   * Plasma glucose levels greater than 200 mg/dL 2 hours after OGT
   * Casual plasma glucose greater than 200 mg/dL combined with diabetic symptoms.
2. Endothelial dysfunction defined by FMD <4%
3. No changes of medication for 2 months
4. Significant PAOD (level IIb, III)

Exclusion Criteria:

1. Ejection fraction <30%
2. Malignoms
3. Terminal renal failure with hemodialysis
4. Relevant cardiac arrhythmias
5. Acute inflammation defined as CRP >0,5 mg/dl
6. PAOD (level IV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-10; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Vascular function | before treatment and after 30 and 60 days

SECONDARY OUTCOMES:
pain free walking distance | before treatment and 30 and 60 days afterwards

CONTACTS AND LOCATIONS:
Overall Officials: Tienush Rassaf, MD, Principal Investigator — Clinic for Cardiology, University Düsseldorf
Locations (1):
- Heinrich-Heine-University, Düsseldorf, Düsseldorf, Germany